CLINICAL TRIAL: NCT06616753
Title: Evaluation of Patients' Knowledge of Their Vaccination Status and Their Relationship to Vaccination at Melun Hospital : Observational Trial
Brief Title: Evaluation of Patients' Knowledge of Their Vaccination Status and Their Relationship to Vaccination at Melun Hospital
Acronym: StatutvaxPat
Status: Recruiting | Type: Observational
Sponsor: Groupe Hospitalier Sud Ile-de-France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01028-37
Record Dates: First submitted 2023-12-15; First posted 2024-09-27 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-09

CONDITIONS: Vaccinia
MeSH Terms: conditions — Vaccinia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: vaccination status — knowledge of own vaccination status

SUMMARY:
The goal of this observational study is to learn about the rate of knowledge of own vaccination status among patients hospitalized at Melun hospital. The main questions it aims to answer are:

* the rate of knowledge of its vaccination status among patients hospitalized at Melun hospital
* hospitalized patients' attitude to vaccination in general. Evaluate the number of patients wishing to update their vaccination status. Observe the influence of various factors (gender, occupation, presence or absence of GP, chronic illness) on vaccination status in Melun, France Participants will be asked to complete a questionnaire during hospitalization.

DETAILED DESCRIPTION:
As part of the national "European Vaccination Week" event organized by the French Ministry of Health and Prevention, we are asking a sample of patients hospitalized in our hospital to complete a questionnaire on their knowledge of their vaccination status, and to assess their relationship with vaccination.

Questionnaire administered to patient during hospitalization (n=140 patients). Patients randomly selected by the Department of Medical Information of the hospital at the beginning of the survey week.

Patients randomly selected from each of the 10 departments of the CH of Melun (internal medicine, infectious diseases, gastroenterology, pneumology, surgery, BCR medicine, cardiology, nephrology, follow-up care and rehabilitation and geriatrics) and accompanied to complete a questionnaire set up by the Public Health Unit (USP) and Hygiene Operational Team (EOH) of the CH of Melun.

ELIGIBILITY:
Inclusion Criteria :

* French-speaking and non-demented patient : able to speak and understand French and without dementia
* Adult patient (Age ≥ 18 years)
* Main place of residence in France
* Hospitalized in a department of the CH of Melun

Exclusion Criteria :

* Does not speak French or dementia
* Patient's refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at CH Melun
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of knowledge of own vaccination status | Day 1

SECONDARY OUTCOMES:
Evaluate the number of patients wishing to update their vaccination status | Day 1
3.Observe the influence of various factors in vaccination status at Melun Hospital : 3.1 % of each gender 3.2 % of patients with a specefic occupation 3.3 % of patients with or without a treating physician 3.4 Rate of patients with chronic illness | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: CORALIE NOEL, Principal Investigator — Groupe Hospitalier Sud Ile-de-France
Locations (1):
- Groupe Hospitalier Sud Ïle de France, Melun, Seine Et Marne, France

DOCUMENTS (1):
  • Study Protocol (2023-09-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT06616753/Prot_000.pdf